CLINICAL TRIAL: NCT06426511
Title: Consolidation Toripalimab Therapy Guided by Circulating Tumor DNA (ctDNA)-Minimal Residual Disease (MRD) for Completely Resected Stage IB-IIIA Non-small-cell Lung Cancer (Without EGFR or ALK Alterations for Nonsquamous Lung Cancer)
Brief Title: ctDNA-MRD Guided Consolidation Toripalimab in Stage IB-IIIA NSCLC
Acronym: CONTINUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO10112
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Incorporate ctDNA-MRD to personalize the administration of consolidation toripalimab therapy for completely resected stage IB-IIIA NSCLC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation for undetectable ctDNA after adjuvant therapy (Experimental): Observation follow-up for patients with undetectable ctDNA after 4 cycles of adjuvant chemotherapy plus toripalimab.
  Interventions: Drug: Toripalimab+Chemotherapy
- Consolidation toripalimab for detectable ctDNA after adjuvant therapy (Active Comparator): Consolidation toripalimab therapy for up to 13 cycles for patients with detectable ctDNA after 4 cycles of adjuvant chemotherapy plus toripalimab.
  Interventions: Drug: Toripalimab+Chemotherapy followed by consolidation toripalimab

INTERVENTIONS:
Drug: Toripalimab+Chemotherapy — After surgical resection, patients received 4 cycle of toripalimab (240 mg) in combination with platinum-based adjuvant treatment. Administration of standard postoperative adjuvant chemotherapy for stage IB disease was not mandatory; decisions about whether patients with IB disease would receive adjuvant chemotherapy were made by the physicians.
  Arms: Observation for undetectable ctDNA after adjuvant therapy
Drug: Toripalimab+Chemotherapy followed by consolidation toripalimab — After surgical resection, patients received 4 cycle of toripalimab (240 mg) in combination with platinum-based adjuvant treatment, and then maintenance treatment with single-agent toripalimab (240 mg) once every 3 weeks for up to 13 cycles.
  Administration of standard postoperative adjuvant chemotherapy for stage IB disease was not mandatory; decisions about whether patients with IB disease would receive adjuvant chemotherapy were made by the physicians.
  Arms: Consolidation toripalimab for detectable ctDNA after adjuvant therapy

SUMMARY:
This study aims to incorporate circulating tumor DNA (ctDNA)-minimal residual disease (MRD) to personalize the administration of consolidation toripalimab therapy in resected stage IB-IIIA non-small-cell lung cancer (NSCLC) after adjuvant therapy. Toripalimab is a humanized monoclonal antibody for human programmed cell death protein 1. Toripalimab was approved as a consolidation treatment after perioperative therapy in combination with chemotherapy for resectable stage III NSCLC.

DETAILED DESCRIPTION:
Most patients with stage IB-IIIA non-small cell lung cancer (NSCLC) are managed with surgery, follow by standard-of-care adjuvant platinum-based chemotherapy. However, postoperative recurrence rates remain high. Recent years, the role of checkpoint inhibitors has been proven to be effective in patients with advanced NSCLC, and even in patients with resectable NSCLC. Emerging data supports the use of consolidation checkpoint inhibitors therapy in localized NSCLC. Based on the results from Neotorch trial, consolidation toripalimab therapy led to a significant improvement in event-free survival for patients with resectable NSCLC. However, not all patients may benefit from consolidation therapy. Circulating tumor DNA (ctDNA) has emerged as a promising biomarker for early detection of minimal residual disease (MRD) in cancer surveillance. There is a critical need to identify MRD after curative therapies to determine which patients may benefit from consolidation toripalimab therapy. The aim of this study is to explore whether observation follow-up for patients with negative ctDNA after adjuvant therapy has a non-inferior prognosis for patients with positive ctDNA and received consolidation toripalimab therapy. This study aims to incorporate ctDNA-MRD to personalize the administration of consolidation toripalimab therapy for completely resected stage IB-IIIA NSCLC (without EGFR or ALK alterations for nonsquamous NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have undergone complete surgical resection (R0) of their stage IB , II and select IIIA NSCLC according to the AJCC 8th edition staging;
* Squamous or non-squamous NSCLC histology;
* Subjects should be without EGFR or ALK alterations for nonsquamous NSCLC;
* Male and female, aged 18-75 years;
* Surgery for lung cancer must be completed ≤ 60 days prior to study treatment;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level);
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN;
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min;
* Female subjects should not be pregnant or breast-feeding;
* Written informed consent provided. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study.

Exclusion Criteria:

* Not R0 resection, or metastatic disease.
* Subjects with known EGFR sensitive mutations or ALK translocation, EGFR and ALK mutation status needs to be identified for the subjects with non-squamous NSCLC;
* Previous treatment with systemic antitumor therapy for NSCLC;
* Severe allergic reaction to other monoclonal antibodies;
* Subjects with any known or suspected autoimmune disorder or immunodeficiency, with the following exceptions: hypothyroidism, hormone therapy is not needed, or well controlled at physiological dose; controlled type I diabetes;
* Uncontrolled active hepatitis B (defined as positive hepatitis B surface antigen in screening period with HBV-DNA detected higher than the upper limit of normal at the clinical laboratory of the study center); active hepatitis C (defined as positive hepatitis C surface antibody in screening period and positive HCV-RNA);
* Vaccination of live vaccine within 30 days prior to the first dose;
* Evidence of clinically active interstitial lung disease;
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Inability to comply with protocol or study procedures;
* Any unstable systemic disease (including active infection, active tuberculosis uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease);
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study and may confuse the study results;
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Women who are pregnant or nursing.
* Ingredients mixed with small cell lung cancer patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The 2-year DFS rate of ctDNA-MRD guided consolidation toripalimab | Baseline to 24 months
  Determine if ctDNA-MRD guided consolidation toripalimab has a non-inferior 2-year DFS to direct 13 cycles of consolidation toripalimab therapy.
  2-year DFS was defined as the proportion of patients who were disease free at 2 years.

SECONDARY OUTCOMES:
The 2-year OS rate of ctDNA-MRD guided consolidation toripalimab | Baseline to 24 months
  Determine if ctDNA-MRD guided consolidation toripalimab has a non-inferior 2-year OS to direct 13 cycles of consolidation toripalimab therapy.
  2-year OS was defined as the proportion of patients who were alive at 2 years.
The 2-year DFS in patients with persistently detectable ctDNA | Baseline to 24 months
  Estimate the 2-year DFS in patients with persistently detectable ctDNA after receiving ≥6 months of consolidation toripalimab.
Percentage of patients with undetectable ctDNA after consolidation toripalimab. | Baseline to 15 months
  Percentage of patients with undetectable ctDNA after consolidation toripalimab of 13 cycles.
Percentage of patients with detectable ctDNA after adjuvant chemotherapy plus toripalimab. | Baseline to 3 months
  Percentage of patients with detectable ctDNA after 4 cycles of adjuvant chemotherapy plus toripalimab.
Adverse Events | Baseline to 36 months
  Adverse Events were monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP